CLINICAL TRIAL: NCT07053917
Title: Psychedelic Healing: Adjunct Therapy Harnessing Opened Malleability
Acronym: PHATHOM
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Rose Hill (Unknown); Usona Institute (Other); University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00274773
Record Dates: First submitted 2025-05-30; First posted 2025-07-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Chronic Stroke; Intracerebral Haemorrhage; Intracerebral Haemorrhage (ICH); Intracerebral Hemorrhage Basal Ganglia; Ischemic Stroke; Ischemic Stroke and Hemorrhagic Stroke; Hemiparesis After Stroke; Hemiplegia Following Ischemic Stroke; Hemiplegia and Hemiparesis; Hemiplegia and/or Hemiparesis Following Stroke; Middle Cerebral Artery Stroke
Keywords: psychedelic; stroke; chronic stroke; intracerebral hemorrhage; stroke recovery; motor recovery; poststroke recovery; poststroke motor recovery; hemiparesis recovery; psychedelic safety
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage; Ischemic Stroke; Hemorrhagic Stroke; Hemiplegia; Paresis; Infarction, Middle Cerebral Artery | interventions — Psilocybin

STUDY DESIGN:
Masking Description: Phase 1 safety trial requires no blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 25 mg of psilocybin (Experimental): Participants will receive 25 mg of psilocybin
  Interventions: Drug: Psilocybin (Usona Institute)
- 12.5 mg + 12.5 mg of psilocybin (Experimental): Participants will receive 12.5 mg of psilocybin followed by another 12.5 mg of psilocybin 2 hours after the first dose.
  Interventions: Drug: Psilocybin (Usona Institute)

INTERVENTIONS:
Drug: Psilocybin (Usona Institute) — Participants will receive psilocybin to test its safety. Secondary outcomes will assess recovery from post-stroke deficits.

SUMMARY:
The main purpose of the current studies is to evaluate the safety and tolerability of psilocybin in patients with chronic stroke.

DETAILED DESCRIPTION:
Stroke is the leading cause of death and adult disability worldwide, and every year more than 795,000 people in the United States have a stroke. According to the National Stroke Association, only 10 percent of people who have a stroke recover completely, while 50 percent experience moderate to severe long-term disability, including significant impairment in language, cognition, motor, and sensory skills, which require special care or long-term care in a nursing home or other facility. Therefore, in the United States alone, nearly 400,000 people per year will suffer the lasting debilitating consequences of stroke. Previous studies have indicated that rehabilitation following stroke is constrained by a so-called 'critical' or 'sensitive' period. While this learning window can be extended or enhanced, once the post-stroke rehabilitation critical period has closed, clinically applicable manipulations that can reopen it are lacking.

Recently the investigators have shown that the psychedelic compounds like psilocybin, lysergic acid diethylamide (LSD), and 3,4-methylenedioxmethamphetamine (MDMA) can reopen a novel critical period for social reward learning. The adage "you can't teach an old dog new tricks" captures a certain truth about the brain. Specifically, a young person's brain is much more malleable (e.g., able to make new motor-memories and store new motor-memories) compared to an adult's brain. Neuroscientists call these periods of heightened sensitivity to input "critical periods." Based on these observations the investigators posit that psychedelic compounds serve as the long sought-after "master key" for unlocking critical periods across the brain. Ongoing preclinical studies are examining this possibility, with the goal of determining the therapeutic potential of psychedelics (including psilocybin) as adjunct therapies for any intervention whose clinical efficacy may be constrained by critical period closure, including post-stroke rehabilitation.

The main purpose of the proposed studies is to evaluate the safety and tolerability of psilocybin in stroke patients (Phase 1). as a secondary aim the investigators will collect data on the efficacy of psilocybin in effecting motor recovery in post-stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Over age 18 years, inclusive.
* Ischemic or hemorrhagic stroke confirmed by CT or MRI, at least 12 months prior to admission date
* Ability to give informed consent and understand the tasks involved.
* Agree that, for the study duration, will refrain from: (1) No new prescription medications during the time of the study without approval of the study team, (2) taking any herbal supplement (except with prior approval of the research team), (3) taking any nonprescription medications with the exception of: 1. non-steroidal anti-inflammatory drugs. 2. acetaminophen. 3. vitamins. 4. or other over-the-counter medications approved by the research team
* Are willing to follow restrictions and guidelines concerning medications, consumption of food, beverages, and nicotine the night before and just prior to psilocybin administration.
* Agree to have transportation other than driving themselves home or to where the participants are staying after the administration of psilocybin.
* Are willing to be contacted via telephone for all necessary telephone contacts.
* Must have a negative pregnancy test if able to bear children.
* Must provide a contact (relative, spouse, close friend or other caregiver) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal.
* Must agree to inform the investigators within 48 hours of any new medical conditions and procedures.
* Are proficient in speaking and reading English.
* Agree to have all clinical visit sessions recorded to audio and video.
* Agree to not participate in any other interventional clinical trials during the duration of this study.

Exclusion Criteria:

* Taking one of the following medications in the 30 days prior to psilocybin administration:

  1. selective serotonin reuptake inhibitor (SSRI)
  2. Serotonin-norepinephrine reuptake inhibitors (SNRI)
  3. Buproprion
  4. Valproic acid
  5. Zolpidem
  6. Trazodone
  7. Carbamazepine.
  8. tricyclic antidepressants
  9. Monoamine Oxidase Inhibitors
  10. Mirtazapine

  l. Lithium m. Buspirone n. Atypical antipsychotics o. Zolpidem p.Carbamazepine q. Clonazepam r. Gabapentin s. Lamotrigine t. Levetiracetam u. Phenobarbital v. Phenytoin w. Topiramate x. Valproic Acid y. Zonisamide
* History of medically significant suicide attempt.
* Evidence of acute cardiac dysfunction as evidenced by either elevated troponin or EKG changes within 48 hours of administration.
* Systolic blood pressure that is greater than 150 mmHg systolic on > 2 readings during the 7-day monitoring period AND blood pressure medication management has been assured.
* Diastolic blood pressure that is greater than 100 mmHg systolic on > 2 readings during the 7-day monitoring period AND blood pressure medication management has been assured.
* Systolic blood pressure is less than 90 mmHg systolic on > 2 readings during the 7-day monitoring period after blood pressure medication management has been assured.
* Diastolic blood pressure is less than 30 mmHg systolic on > 2 readings during the 7-day monitoring period after blood pressure medication management has been assured.
* Systolic blood pressure exceeds 160 mmHg or is less than 90 mmHg immediately prior to administration of psilocybin; patients are allowed to be on anti-hypertensives.
* Diastolic blood pressure exceeds 100 mmHg or is less than 30 mmHg immediately prior to administration of psilocybin; patients are allowed to be on anti-hypertensives.
* Cognitive impairment that, in the estimation of the study team, would preclude the use of the MindPod Dolphin.
* History of physical or neurological condition that interferes with study procedures or assessment of motor function (e.g. severe arthritis, severe neuropathy, Parkinson's disease).
* Social and/or personal circumstances that interfere with ability to perform follow up assessments.
* Are pregnant or nursing.
* Weigh less than 48 kg.
* Are not able to give adequate informed consent.
* Are actively abusing opioids, cocaine, Phencyclidine (PCP), amphetamines, or alcohol.
* Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (SCID-5) criteria for moderate or severe substance use disorder
* Diagnosis of schizophrenia, history of prior psychosis, anxiety requiring hospitalization, or Type 1 bipolar.
* Hypernatremia
* Hypokalemia (but can have received repletion during the prior 24 hours)
* Hyperkalemia
* Glomerular filtration rate of < 30 ml/min
* Elevated of white blood cell count
* Hemoglobin < 7 g/dl
* Platelet count < 100,000 g/dl
* Acute cardiac dysfunction demonstrated by either troponin elevation (chronic elevation is acceptable), or EKG changes suggestive of acute coronary syndrome.
* Active suicidal ideation as assess by the C-SSRS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Stability of systolic and diastolic blood pressure (mmHg) | up to 24 hours post-psilocybin administration
  Will be measuring the number of participants that meet these criteria:
  1. no sustained elevation of systolic blood pressure of more than 180 mmHg on more than two readings sustained for more than 20 minutes.
  2. no sustained elevation of diastolic blood pressure of more that 120 mmHg on more than two reading sustained for more than 20 minutes.
  3. No sustained reduction of systolic blood pressure of less than 70 mmHg on more than two readings sustained for more than 20 minutes.
  4. No sustained reduction of diastolic blood pressure of less than 40 mmHg on more than two readings sustained for more than 20 minutes

SECONDARY OUTCOMES:
Number of adverse changes in vital signs that require medical attention | up to 24 hours post-psilocybin administration
  Adverse change in vital signs, not otherwise meeting specified outcome criteria, that a treating provider feels requires medical intervention.
Number of changes in psychiatric symptoms that require medical intervention | up to 24 hours post-psilocybin administration
  Significant psychiatric symptoms within 24 hours post-dosing as determined by clinical staff to require medical intervention
Stability of pulse assessed by heart rate monitoring | up to 24 hours post-psilocybin administration
  no resting tachycardia for more than 20 minutes defined as heart rate greater than 110 bpm, or resting bradycardia for more than 20 minutes defined as less than 40 bpm.
Oxygen Percent Saturation | up to 24 hours post-psilocybin administration
  Stability of pulse oximetry. No reduction of percent saturation of less than 87% as assess by pulse oximetry on more than two readings sustained for more than 10 minutes.
Number of participants with no change in EKG suggestive of ischemia | up to 24 hours post-psilocybin administration
  No change in EKG suggestive of ischemia
Number of participants without seizures | up to 24 hours post-psilocybin administration
  No seizures assessed by clinical observation and examination
Number of Participants without elevation of cardiac troponin | up to 24 hours post-psilocybin administration
  Troponin assessed by serum quantification
Suicidal ideation assessed by Columbia Suicide Severity Rating Scale (C-SSRS) | Day 1, prior to dosing-24 hours post-dosing (+/- 5 hours) weekly, up to 3 weeks
  Suicidal ideation as assessed by the Columbia Suicide Severity Rating Scale (C- SSRS) before, during and after experimental sessions and on selected days of telephone or face-to-face contact. Score range 0-25 with higher scores indicating more severe suicidal ideation.
Number of deviations from pre-dosing electrolyte levels as assessed by CMP | Pre-dosing and between 8 and 24 hours post-psilocybin dosing
  Deviation from pre-dosing values of sodium, potassium, chlorine, and calcium, will be assessed by comprehensive metabolic panel (CMP)
Neurologic Impairment as assessed by The National Institutes of Health Stroke Scale (NIHSS) | 30 days and 90 days
  Secondary recovery outcome. Scores range from 0 to 42, with higher scores indicating increasing severity
Motor Function as assessed by the Fugl-Meyer Upper Extremity Motor Assessment (FM-UE) | 30 days and 90 days
  Secondary recovery outcome. The score range is 0 to 66. A lower score indicates impaired motor function in the upper extremity assessed.
Amount of recovery of arm-hand function as assessed by the Action Research Arm Test (ARAT) | 30 days and 90 days
  Secondary recovery outcome. Scores range from 0-to-57 with a higher score indicating a better outcome.
Global disability as assessed by the Modified Rankin Scales (mRS) | 30 days and 90 days
  Secondary recovery outcome. Modified Rankin Scales (mRS) is a measure of global disability. Total Scale range is 0-6, with lower values indicating better outcomes.
Function as assessed by the Barthel Index (BI) | 30 days and 90 days
  Secondary recovery outcome. Barthel Index scores range from 0 to 100, with higher scores indicating greater levels of function.
Montreal cognitive assessment (MOCA) | 30 days and 90 days
  Secondary recovery outcome. MOCA score ranges from 0-30, with higher score being better performance.
Digital hand kinematics | 30 days and 90 days
  Secondary recovery outcome. Change in fingertip individuation index as assessed by kinematic measurement of digit movement using a device that uses sensor-based technology to capture joint range of motion. Full extension and flexion of each digit in isolation will be captured using this technology and compared.
Change in finger dexterity as assessed by the nine-hole peg test (9PHT) | 30 days and 90 days
  Secondary recovery outcome. The Nine-Hole Peg Test (9HPT) is used to measure finger dexterity in patients with various neurological diagnoses. Participants are asked to place pegs into the holes one at a time, then remove them one at a time, and place them back in the container as fast as they can.
Grasp Performance | 30 and 90 days
  Secondary recovery outcome. Change in gross grasp will be measured using dynamometry in pours of force output. three measure will be take on the right and left hand and the value will be averaged using a calibrated dynamometer. greater force output is equal to greater grip strength.
10m walk time | 30 days and 90 days
  Secondary Recovery Outcome. Patients are asked to walk 10m. faster is better.
Depression as assessed by the Patient Health Questionnaire (PHQ) | 30 days and 90 days
  Secondary recovery outcome. Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe (range of 0-27)
Stroke Impact Scale (SIS)-16 | 90 days
  The Stroke Impact Scale (SIS)-16 consists of 16 items from the 4 physical domains (strength, hand function, mobility, and ADL/IADL) to assess recovery post-stroke. Total score ranges between 0-100; higher scores are better.
Secondary recovery outcome - post-study assessment survey | 90 days
  Survey designed to assay participant's enjoyment and self-assessed recovery

CONTACTS AND LOCATIONS:
Overall Officials: Victor Urrutia, M.D., Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No